CLINICAL TRIAL: NCT02921165
Title: Comparison of Topical Analgesic With Saline Rinses in Post Extraction Healing Among Hypertensive and Non-hypertensive Subjects
Brief Title: Comparison of Topical Analgesic With Saline Rinses in Post Extraction Healing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Rabia Ali, Dr. Rabia Ali, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AgaKhanUniversity
Record Dates: First submitted 2016-09-23; First posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Periodontitis; Dental Caries; Hypertension
Keywords: tooth extraction; tooth socket healing; hypertension; rinses
MeSH Terms: conditions — Periodontitis; Dental Caries; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Non hypertensive Intervention: On analgesic mouth rinses (dissolved Aspirin)
  Interventions: Drug: analgesic mouth rinses (dissolved Aspirin)
- Group 2 (Experimental): Hypertensive Intervention: On analgesic mouth rinses (dissolved Aspirin)
  Interventions: Drug: analgesic mouth rinses (dissolved Aspirin)
- Group 3 (Experimental): Non Hypertensive Intervention: On normal saline rinses.
  Interventions: Drug: Normal saline rinses.

INTERVENTIONS:
Drug: analgesic mouth rinses (dissolved Aspirin) — Group 1 and Group 2 patients will be prescribed analgesic mouth rinses (dissolved Aspirin) twice daily along with the standard prescription of analgesics and antibiotics.
  Other Names: water dissolved aspirin rinse
  Arms: Group 1; Group 2
Drug: Normal saline rinses. — Non Hypertensive patients will be prescribed normal saline rinses twice daily along with the standard prescription of analgesics and antibiotics.
  Other Names: warm saline rinses; salt water rinses
  Arms: Group 3

SUMMARY:
The aim of this study is to determine the beneficial effect of mouth rinses, both topical analgesic and saline regimens as an adjuvant therapy in the presence of standard prescription of post-operative pain killers on the progress of socket healing following routine dental extraction.

DETAILED DESCRIPTION:
Hypertension is a highly prevalent cardiovascular disease, which affects over 1 billion people worldwide. It varies with age, race, education and so forth.1 The National Health Survey of Pakistan estimated that hypertension affects 18% of adults and 33% of adults are above 45 years old.2It is a common disease encountered in dental setting. Its wide spreading, terrible consequences, and life-long treatment require an attentive approach by dentists. Knowledge of hypertension is important for dentists especially for risk assessment for dental treatment. This may lead to improved monitoring and treatment.

Dental treatment in hypertensive patients necessitates special attention, because any stressful procedure may increase blood pressure and trigger acute complications such as cardiac arrest or stroke. Extractions are usually done for teeth which are not salvageable. Dentists routinely advice use of warm saline rinses to help in healing of post extraction socket. But for hypertensive patients this recommendation is potentially harmful There is no evidence based guidelines on using saline rinses for post extraction oral care among hypertensives. Moreover, advantage of orally dissolved topical analgesics in addition to orally administered analgesic is questionable.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects requiring simple tooth extraction (elevator or forceps) which were either known cases of controlled hypertension under medical treatment or confirmed non hypertensives.

Exclusion Criteria:

* Subjects requiring surgical tooth extraction involving bone removal and suturing, uncontrolled systemic disorders (diabetes mellitus, hypertension, blood coagulopathies, metabolic bone disorders), on platelet aggregation therapy or warfarin (anticoagulants) or bisphosphonate therapy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with unhealed extraction socket | Number of participants with unhealed extraction socket at 7th day

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ali, BDS, Principal Investigator — Aga Khan University; Farhan Raza Kahn, FCPS, Study Director — Aga Khan University

IPD SHARING:
Plan to Share IPD: No